CLINICAL TRIAL: NCT02674919
Title: The Efficacy of a 10-week Intervention, Using the Nordic Hamstring Exercise, on Repeated-sprint Ability in Football (Soccer) Players - a Randomized Controlled Trial
Brief Title: Nordic Hamstring and Repeated-sprint Ability in Football (Soccer) Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Aspetar (Other)
Responsible Party: Principal Investigator, Lasse Ishøi, PT, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NHE-2016-LI
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Repeated-sprint Ability
Keywords: Repeated-sprint ability; Nordic Hamstring exercise; Eccentric hamstring muscle strength

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nordic Hamstring (Experimental): The Nordic Hamstring group performs a progressive strengthening program (Mjolsnes et al., 2004) comprising of the Nordic Hamstring exercise during a period of 10 weeks. The training load increases from one session per week in week 1 to 3 sessions per week in week 3-10. Number of sets and repetitions progressively increase from 2 to 3 and 5 to 12, respectively. The exercise program is performed in the end of a regular football training session.
  Interventions: Other: Nordic Hamstring
- Control (Other): The control group are asked not to perform the exercise or any other specific strength training for the hamstring muscles and to continue to play football as usual.
  Interventions: Other: Control

INTERVENTIONS:
Other: Nordic Hamstring
  Other Names: Hamstring lowers; Nordic lowers; Hamstring Curl
  Arms: Nordic Hamstring
Other: Control
  Arms: Control

SUMMARY:
The purpose of the study is to investigate the efficacy of a 10-week intervention, using the Nordic Hamstring exercise, on repeated-sprint ability in male sub-elite football players. The primary outcome measure is total sprint time during 4x6 sprint of 10 meters measured using dual-beam photoelectric cells. Additionally, eccentric knee flexor strength is measured using the Nordbord hamstring strength measure. The hypothesis is that strength training of the knee flexor muscles elicited by the Nordic Hamstring exercise will result in enhanced repetitive sprint-ability expressed as a decrease in total sprint time. Furthermore, baseline data is used to assess to correlation between eccentric hamstring strength and active hamstring flexibility AND sprint performance.

ELIGIBILITY:
Inclusion Criteria:

* Sub-elite Danish football player
* Age 17-35.
* Able to participate fully in competitive football activities at the time of testing

Exclusion Criteria:

* Hamstring pain resulting in loss of training and matches 2 months prior to study initiation.
* Specific systematic strength training of the hamstring muscles (>1/week) in the preceding 2 months before study initiation.
* Specific systematic sprint training (>1/week) in the preceding 2 months before study initiation.
* Longstanding injury (>6 weeks) in the lower extremities in the preceding 6 months to study initiation.

Ages: 17 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Total sprint time measured during 4x6 sprints of 10 meters. The sprints are performed every 15s and the sets are separated by 3 minutes of rest. | Measured prior to and after the intervention period (at week 0 & 10)

SECONDARY OUTCOMES:
Single sprint times (best sprint time, sprint time during last sprint). | Measured prior to and after the intervention period (at week 0 & 10)
Maximal eccentric knee flexor strength measured using Nordbord device | Measured prior to and after the intervention period (at week 0 & 10)
Eccentric knee flexor strength endurance measured during 12 repetitions of the Nordic Hamstring exercise using Nordbord device. | Measured prior to and after the intervention period (at week 0 & 10)
Active range of motion of hamstring muscles measured using inclinometer. | Measured prior to and after the intervention period (at week 0 & 10)
Correlation between eccentric hamstring strength and active hamstring flexibility AND sprint performance. | Measured prior to the intervention (at week 0)

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Ishøi, Principal Investigator — Hvidovre University Hospital. University of Southern Denmark; Per Hölmich, Study Chair — Hvidovre University Hospital. Aspetar; Per Aagaard, Study Chair — University of Southern Denmark; Kristian Thorborg, Study Chair — Hvidovre University Hospital; Thomas Bandholm, Study Chair — Hvidovre University Hospital; Andreas Serner, Study Director — Hvidovre University Hospital. Aspetar
Locations (1):
- Both the intervention and testing included in protocol will be conducted in the facilities of the included football clubs in Copenhagen, Denmark., Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All individual data regarding primary and secondary outcome measures.
Time Frame: Data are available indefinitely at https://www.dropbox.com/s/8g2hve95csz42zp/IPD.xlsx?dl=0
Access Criteria: No access criteria.

REFERENCES:
- [Background] Mjolsnes R, Arnason A, Osthagen T, Raastad T, Bahr R. A 10-week randomized trial comparing eccentric vs. concentric hamstring strength training in well-trained soccer players. Scand J Med Sci Sports. 2004 Oct;14(5):311-7. doi: 10.1046/j.1600-0838.2003.367.x. PMID 15387805
- [Derived] Ishoi L, Holmich P, Aagaard P, Thorborg K, Bandholm T, Serner A. Effects of the Nordic Hamstring exercise on sprint capacity in male football players: a randomized controlled trial. J Sports Sci. 2018 Jul;36(14):1663-1672. doi: 10.1080/02640414.2017.1409609. Epub 2017 Dec 1. PMID 29192837